CLINICAL TRIAL: NCT02791386
Title: Rescue Treatment Pattern, Drug Resistance Recurrence, and Direct Medical Costs Associated With Chinese Patients With Chronic Hepatitis B and Drug Resistance to Nucleot(s)Ide Analogue Monotherapy: A Retrospective Cohort Study
Brief Title: Rescue Treatment Pattern, Drug Resistance Recurrence, and Direct Medical Costs Associated With Chinese Patients With Chronic Hepatitis B and Drug Resistance to Nucleot(s)Ide Analogue Therapy
Acronym: NAs resistance
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-508
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chinese Patients With CHB and Drug Resistance to NA Therapy

SUMMARY:
The purpose of this study is to describe current rescue treatment pattern for nucleot(s)ide analogue (NA) resistance and assess the real-world treatment outcomes and health resources utilization of rescue treatments for drug resistance in a clinical cohort of Chinese patients with chronic hepatitis B (CHB).

ELIGIBILITY:
Inclusion Criteria:

* CHB patient with drug resistance confirmed by hepatitis B virus (HBV) gene mutation and virological breakthrough
* Patient receiving rescue treatments for drug resistance to previous NA therapy for CHB
* Patient who was regularly followed at least every 6 months for drug resistance at the tertiary liver clinic of SXH

Exclusion Criteria:

* Patient with a diagnosis of hepatocellular carcinoma, decompensated cirrhosis, and/or liver transplantation prior to the development of drug resistance to NA therapy for CHB
* Patient with co-infection with hepatitis C virus, hepatitis D virus, and/or human immunodeficiency virus
* Patient with life expectancy less than 6 months after the date of the first laboratory test indicating drug resistance

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Direct medical costs associated with CHB patients who were regularly followed for drug resistance to NA therapy at the tertiary liver clinic of the Second Xiangya Hospital (SXH) in Changsha, Hunan, China | Retrospectively collected from March 31, 2008 to August 15, 2016
Rescue treatments effect on direct medical costs associated with CHB patients who were followed for drug resistance to NA therapy at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016

SECONDARY OUTCOMES:
Rescue treatment patterns associated with CHB patients who were regularly followed for their drug resistance to NA therapy at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016
Virological response recurrence associated with rescue treatments for drug resistance to NA therapy in CHB patients who were followed at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016
Biochemical response recurrence associated with rescue treatments for drug resistance to NA therapy in CHB patients who were followed at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016
Drug resistance recurrence associated with rescue treatments for drug resistance to NA therapy in CHB patients who were followed at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016
Rescue treatments effect on liver-related complications in CHB patients who were followed up for drug resistance to NA therapy at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016
Rescue treatments effect on mortality in CHB patients who were followed up for drug resistance to NA therapy at the tertiary liver clinic of SXH | Retrospectively collected from March 31, 2008 to August 15, 2016

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Changsha, Hunan, China

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx